CLINICAL TRIAL: NCT02239796
Title: A Feasibility Study for a Randomised Controlled Trial of Transcutaneous Posterior Tibial Nerve Stimulation to Alleviate Stroke-related Urinary Incontinence.
Brief Title: Feasibility Controlled Trial of Tibial Nerve Stimulation for Stroke Related Urinary Incontinence
Acronym: TREAT-UI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glasgow Caledonian University (Other)
Collaborators: The Stroke Association, United Kingdom (Other); University of Central Lancashire (Other); Nursing, Midwifery & Allied Health Professions Research Unit (Unknown); NHS Greater Glasgow and Clyde (Other); NHS Lanarkshire (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TSA 2013/05
Record Dates: First submitted 2014-08-12; First posted 2014-09-15 (Estimated); Last update posted 2016-05-26 (Estimated); Status verified 2016-02

CONDITIONS: Stroke; Urinary Incontinence
Keywords: transcutaneous posterior tibial nerve stimulation; Randomised controlled trial; Feasibility
MeSH Terms: conditions — Stroke; Urinary Incontinence

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- TPTNS (Experimental): 12 stimulation sessions of 30 minutes duration, delivered twice weekly over a 6 week period using a NeuroTrac continence stimulator.
  Two surface electrodes are applied to the non-hemiparetic ankle, where appropriate, or the right ankle where no hemiparesis exists. The electrical stimulator is pre-programmed to safely deliver 30 minutes of continuous stimulation with a pulse frequency of 10 hertz and pulse width 200µs22. The intensity of the current will depend on the stroke survivor's perception threshold and individual comfort and is self-adjusted at each session, but will normally range between 15 and 40 milliamps.
  Interventions: Device: NeuroTrac continence stimulators
- Sham TPTNS (Sham Comparator): The sham stimulation group will self- or carer-deliver a similar programme of twelve, 30 minute sessions twice weekly for 6 weeks NeuroTrac continence stimulator.
  The surface electrodes will be positioned on the lateral malleolar area of the ankle, not the medial aspect, to avoid the posterior tibial nerve.
  The stimulation intensity will be increased until sensation is reported, then turned down to 4mA for the 30 minute session, ensuring that despite avoiding the posterior tibial nerve, there is no therapeutic stimulation provided.
  Interventions: Device: NeuroTrac continence stimulators

INTERVENTIONS:
Device: NeuroTrac continence stimulators — Electrically stimulating the sacral nerve plexus modulates the L4-S3 nerve roots that control bladder function and urethral sphincter activity to eliminate inappropriate detrusor contractions while leaving the micturition reflex intact.
  Transcutaneous posterior tibial nerve stimulation (TPTNS) is a technique of non-invasive retrograde electrical stimulation of the sacral plexus via the sciatic nerve. The posterior tibial nerve, a tributary of the sciatic nerve, is accessed using surface electrodes applied to the medial malleolar area. We are using NeuroTrac continence stimulators.
  Arms: TPTNS
Device: NeuroTrac continence stimulators — We are using NeuroTrac continence stimulators.
  Arms: Sham TPTNS

SUMMARY:
To aim of this study is to establish the feasibility of undertaking a phase III trial of transcutaneous posterior tibial nerve electrical stimulation (TPTNS) to alleviate stroke-related urinary incontinence.

DETAILED DESCRIPTION:
Stroke-related urinary incontinence (UI) persists in more than one third of stroke survivors. It is associated with significant burden including reduced quality of life, increased morbidity and disability. Urgency UI, together with overactive bladder (OAB) symptoms (frequency, urgency, nocturia), is most commonly experienced. Current continence care is limited to lifestyle advice and behavioural interventions such as voiding programmes. There is a reliance on containment approaches and a lack of available options for active treatment. Intermittent electrical stimulation of the posterior tibial nerve (TPTNS) is effective for treating non-stroke neurogenic UI and OAB, but has not been tested in the stroke population. This pilot randomised controlled trial (RCT) aims to test the potential effectiveness of TPTNS for stroke-related bladder dysfunction. Adults with stroke-related UI will be randomised to TPTNS or sham. They and/or their carer will be taught to self-deliver a programme of TPTNS over a six week period. Bladder function, associated healthcare costs and quality of life outcomes will be measured at 6, 12 and 26 weeks. A nested process evaluation will be conducted. Pilot RCT and process evaluation results will inform the design of a phase III RCT of TPTNS to treat urinary incontinence in the stroke population.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged ≥ 18 years, with a diagnosis of stroke based on the WHO criteria (WHO 1989) and stroke-related urinary incontinence of at least once weekly.
* Onset of stroke ≥ 4 weeks previously and discharged from hospital to own home following a new stroke episode within the previous 6 months.
* Physically, cognitively and communicatively able and willing to learn to apply TPTNS or has carer who is able and willing to learn.

Exclusion Criteria:

* Pre-existing urinary incontinence prior to stroke.
* Current Urinary Tract Infection.
* Voiding dysfunction requiring intermittent/indwelling catheterisation.
* Cardiac pacemaker in situ.
* Concurrent neurological diagnosis eg dementia, Multiple Sclerosis, diabetic neuropathy.
* Reduced/absent sensation at electrode placement sites.
* Post-void residual urine volume of > 150ml.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2014-09; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Frequency of reported episodes of urinary incontinence as a measure of effectiveness. | Up to 16 months
  Positive response to International Consultation on Incontinence Questionnaire-Urinary Incontinence Short-Form (ICIQ-UI SF).
  This outcome will be the primary outcome for a future full evaluation trial, should it prove feasible.

SECONDARY OUTCOMES:
Changes in the severity of urinary incontinence episodes experienced. | Up to 16 months
Number of participants with adverse events as a measure of safety and tolerability. | Up to 16 months
Changes in severity of urinary urgency, frequency and nocturia. | Up to 16 months
  By completion of AUASI
Urinary symptoms experienced on the American Urological Association Symptom Index | Up to 16 months
Mean Urgency Perception Scores recorded on a 3 day bladder diary | Up to 16 months
Patient Perception of Bladder Condition | Up to 16 months
Severity of bowel symptoms | Up to 16 months
Patient Perception of Bowel Condition | up to 16 months
Changes in post-void residual urine volume. | Up to 16 months
Amount of urine leakage in 24 hours | Up to 16 months
Participants perception of independence from any help with activities of daily living | Up to 16 months
  Measured by completion of the Barthel Index Score and Modified Rankin Score.

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Booth, Principal Investigator — Glasgow Caledonian University
Locations (2):
- United Kingdom (2):
  - NHS Ayrshire and Arran, Ayrshire
  - NHS Lanarkshire, Glasgow